CLINICAL TRIAL: NCT06737328
Title: SPiT-frequency I_Peri-implant Mucositis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Odd Carsten Koldsland, Associate Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPiT-frequency I_Peri-implant; REK790097 (Other: Regional Ethic Committee, South East Norway)
Record Dates: First submitted 2024-11-25; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Peri-Implantitis and Peri-implant Mucositis
Keywords: Peri-implant mucositis; Supportive peri-implant treatment; Frequency
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test. Increased treatment frequency (Experimental): Submucosal instrumentation will be performed at baseline, 3 weeks, 6 weeks, 9 weeks, 12 weeks, 16 weeks, 24 weeks and 36 weeks.
  Interventions: Procedure: Submocosal instrumentation using a ultrasonic device (PEEK). Submucosal cleaning
- Control. Conventional frequency (Active Comparator): Submucosal instrumentation will be performed at baseline, 12 weeks, 24 weeks and 36 weeks
  Interventions: Procedure: Submocosal instrumentation using a ultrasonic device (PEEK). Submucosal cleaning

INTERVENTIONS:
Procedure: Submocosal instrumentation using a ultrasonic device (PEEK). Submucosal cleaning — The treatment under study is professional non-surgical, submucosal debridement with ultrasonic instruments with PolyEther Ether Ketone (PEEK) tip followed by copious irrigation with sterile saline

SUMMARY:
This is an interventional clinical study on the peri-implant treatment necessary to improve the clinical conditions surrounding dental implants registered with peri-implant inflammation. The focus of this double-armed, examiner blinded, controlled, randomized clinical trial is to examine the effect of short-term increased frequency of a SPiT (supportive peri-implant treatment) protocol on implants diagnosed with peri-implant mucositis.

The study is a part of a project assessing the frequency of supportive peri-implant therapy. The current is on treatment of peri-implant mucositis (inflammation and no attachment loss at the implants) and secondary prevention of peri-implant mucositis. The other study is a RCT on non-surgical treatment of peri-implantitis (inflammation and exposed implant surface) (REK 790240). Exposure of rough surface may dramatically change the frequency of maintenance needed to improve the inflammatory condition. Thus, a segregation between adequate and low bone level at the implant is necessary.

Subjects with more than one implant and both diagnoses, may be enrolled in both studies, following the frequency of treatment randomized in the peri-implant mucositis study.

DETAILED DESCRIPTION:
At the screening visit, the following tests and examination will be carried out to screen eligible subjects and provide baseline information for those patients that meet the study criteria:

* Anamnestic information as described in the regular electronic dental journal at the Faculty of Dentistry is collected
* Assessment of clinical registrations; suppuration, plaque, gingival bleeding, PPD, Bleeding index score and presence of keratinized mucosa
* Assessment of existing radiographs to ensure the subject and implants are eligible according to inclusion criteria
* Written and oral information on the study will be given
* Thorough information and instruction in plaque control with tools deemed appropriate by the operator
* Information about the study is given orally and written together with informed consent sheet

Visit 1 Baseline Signed inform consent is collected

An experienced, calibrated and board certified specialist in periodontology ("Examiner") performs the following clinical registrations at six sites (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) of the included implants:

Plaque: the presence or absence recognized by running a probe across the marginal surface of the implant (Mombelli et al. 1987). If plaque is present at the implants to be included, oral hygiene instructions are repeated and Baseline examination is rescheduled PICF (peri implant cravicular fluid): Peri-implant crevicular fluid (PICF) will be collected from one site per implant, at the site with the most severe lesion at the baseline Suppuration: the presence or absence after light pressure against gingiva/mucosa or following gentle probing of the peri-implant pocket.

Mucosal bleeding: registered according to the Modified Sulcus Bleeding Index (mBI) (Mombelli et al. 1987).

PPD: recorded with a pressure- sensitive probe (20 g) (University of North Carolina probe, Aesculap, Braun, Tuttlingen, Germany).

Bleeding index score: measured at the implants after probing at six sites, and graded (0-3):

0 = no bleeding,

1. = spot bleeding,
2. = line bleeding
3. = profound bleeding within 30 seconds after measurement of PPD. Presence of keratinized mucosa: registered at the mid buccal site as "adequate" ≥2 mm, "inadequate" <2 mm (Moraschini et al. 2017).

Buccal recession; the distance from a fixed point - suprastructure/abutment connection to the mucosal margin in mm Saliva samples; Stimulated saliva will be collected for 5 min in sterile ice-chilled tubes while chewing on Parafilm.

Immediately after collection, volume of collected saliva will be recorded to determine salivary flow, while pH will be measured using a hand-held pH electrode or pH strips. Buffer capacity will be determined by adding 5 mM HCl in sample of the collect saliva in 3:1 ratio and then measuring the pH with a hand-held pH electrode or pH strips. Remaining saliva will be centrifuged at 7500 × g at 4°C for 10 min and stored in -80°C up to two months prior to further analysis. Total protein content in saliva will be measured using Pierce BCA protein assay, while calcium content will be determined with atomic absorption spectroscopy. Salivary antioxidant activity will be measured using ABTS assay. For these assays, the saliva samples will be thawed immediately prior to analysis and all samples will be discarded immediately after the assay is completed (edited 21.08.23) The following procedures will be performed by "the Operator" Radiographs of the implants showing clear projections of the implant threads at the mesial and distal surfaces will be taken using standard Eggens holders

All included implants receive the following treatment:

Repeated oral hygiene instruction if needed Submucosal instrumentation with ultrasonic device with a PEEK tip followed by copious irrigation with sterile saline Supramucosal polishing using polishing paste and rubber cup Following treatment, if local anesthesia was not applied, the subjects will be asked to grade the level of pain experienced on a 10 cm visual analogue scale (VAS).

The Examiner leaves the room prior to randomization performed by the Operator by opening a concealed envelope stating "test" or "control". Each subject may have more than one implant included in the study. All the implants will be scheduled for the same frequency of SPiT

3-, 6- and 9 weeks following baseline Appointments scheduled for High frequency SPiT implants only. At these time points, all implants are assessed by the Operator (non-blinded examination) and receive supramucosal polishing, submucosal instrumentation as described above and OHI- if necessary VAS scales are registered

12 weeks (3 months) following baseline At this time point, all implants are clinically examined by a blinded Examiner and receive supramucosal polishing as well as submucosal instrumentation and OHI as described above VAS scales are registered

16 weeks (4 months) following baseline Appointments scheduled for High frequency SPiT implants only. At this time points, all implants are assessed by the Operator and receive supramucosal polishing, submucosal instrumentation as described above and OHI- if necessary VAS scales are registered

24 weeks (6 months) following baseline At this time point, all implants are clinically examined by a blinded Examiner and receive supramucosal polishing as well as submucosal instrumentation and OHI as described above by the Operator VAS scales are registered

36 weeks (9 months) following baseline At this time point, all implants are clinically examined by a blinded Examiner and receive supramucosal polishing as well as submucosal instrumentation and OHI as described above by the Operator VAS scales are registered Radiographs are taken according to the baseline examination Referring dentist/dental hygienist (if any) is given written information about the treatment performed and the result, and suggested routines of follow-up is suggested

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 20 years, diagnosed with peri-implant mucositis as defined by the World Workshop 2017 criteria (Berglundh et al., 2018) at an adequate (<0.5mm) bone level Peri-implant mucositis: Bleeding after gentle probing at an implant and no radiographic bone loss)

Exclusion Criteria:

* Previous radiotherapy in the affected area, current use of chemotherapy, systemic long-term corticosteroid treatment.

  * No pregnant or nursing subjects.
  * > class 2 according to the ASA (American Society of Anesthesiologists) physical status classification.
  * HIV positive or other disease severely affecting the immune system
  * If examiners/operators agree the placement of the implant (angle, position, proximity to adjacent implant or tooth) or suprastructure was suboptimal and considered to play a major role in the development of inflammation.
  * Anatomical abnormalities.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-19 (Estimated); Study Completion 2028-01-19 (Estimated)

PRIMARY OUTCOMES:
Peri-implant inflammation | From baseline to 9 months
  To assess the proportion of implants without signs of inflammation (Inflammation is defined as; Bleeding on Probing (BoP) and/or suppuration)

SECONDARY OUTCOMES:
Improvement of inflammation severity | From baseline to 9 months
  Bleeding index (BI) 3, 2, 1, 0 (Roos-Jansåker et al., 2007)

OTHER OUTCOMES:
Extent of inflammation | Baseline to 9 months
  Number of inflamed sites at the implants (0-6)
Reduction of pocket probing depths | Baseline to 9 months
  Pocket depths in mm
Buccal keratinized mucosa | Baseline to 9 months
  Height of keratinized mucosa at the buccal aspect of the implant (in mm)
Progressive bone loss | Baseline to 9 months
  Radiographic changes in bone level at the implant (in mm)
Implant survival | Baseline to 9 months
  Presence of the implant at site, osseointegration intact (mobility grade =0)
Patient related outcome - pain | Baseline to 9 months
  Patient experience of pain in relation to treatment, registered at a VAS-scale 0-100 mm
Accessibility | Baseline to 9 months
  Patient and operators assessment of accessibility for maintenance/treatment, registered as sufficient/insufficient
Sulcus fluid analyses | Baseline to 9 months
  The impact of saliva calcium content, buffer capacity and Ph on the different outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Carl Hjortsjø, Ph.D, Principal Investigator — Institute for Clinical Dentistry, Dental Faculty, University of Oslo
Locations (1):
- Faculty of Dentistry, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publicaton
Access Criteria: Central Contact person and corresponding author of publication